CLINICAL TRIAL: NCT00882752
Title: Retrospective Study Protocol: Report of a New Method Used to Identify the Bacteria Present in a Human Colon Biopsy
Brief Title: Report of a New Method Used to Identify the Bacteria Present in a Human Colon Biopsy Sample
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Principal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-009
Record Dates: First submitted 2008-09-29; First posted 2009-04-16 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Molecular Analysis
Keywords: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — colon biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ulcerative colitius: The method used to identify the microbes in the sample was chosen because it had the potential to provide more exhaustive identification of the bacteria present in the sample as compared to culturing methodology.
  Interventions: Procedure: molecular analysis

INTERVENTIONS:
Procedure: molecular analysis — bowel disease

SUMMARY:
The method used for the biopsy analysis may be able to provide important insights into the complex microbial communities found in the human colon or in complex human infections. Therefore, this methodology may prove useful to other researchers or physicians.

DETAILED DESCRIPTION:
The method used to identify the microbes in the sample was chosen because it had the potential to provide more exhaustive identification of the bacteria present in the sample as compared to culturing methodology. The molecular method worked well, so it is appropriate to share the method with the medical and scientific communities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis
* Age >= 18 years old
* Female

Exclusion Criteria:

Anyone not meeting inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with ulcerative colitis.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The method used for the biopsy analysis may be able to provide important insights into the complex microbial communities found in the human colon or in complex human infections. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Randall Wolcott, MD, Principal Investigator — Southwest Regional Wound Care; Randall Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center